CLINICAL TRIAL: NCT00043277
Title: Pilot Dose Finding And Efficacy Study Of Angiomax® (Bivalirudin) As Primary Anticoagulation In Infants Under Six Months With Thrombosis
Brief Title: Study Of Angiomax In Infants Under Six Months With Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-04
Record Dates: First submitted 2002-08-07; First posted 2002-08-08 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2006-01

CONDITIONS: Thrombosis
Keywords: neonates; thrombosis; bivalirudin; direct thrombin inhibitor
MeSH Terms: conditions — Thrombosis | interventions — bivalirudin

INTERVENTIONS:
Drug: Angiomax (bivalirudin)

SUMMARY:
The goals of this study are:

1. To assess the safety of bivalirudin in infants under six months with arterial or venous thrombosis;
2. To determine the dose of bivalirudin required to achieve adequate anticoagulation as measured by the activated clotting time (ACT) or activated partial thromboplastin time (aPTT) in Infants Under Six Months with arterial or venous thrombosis;
3. To determine the outcome of patients on bivalirudin with respect to thrombus resolution and bleeding complications compared to patients on unfractionated heparin (UH) or low molecular weight heparin (LMWH).

DETAILED DESCRIPTION:
The goals of this study are:

1. To assess the safety of bivalirudin in infants under six months with arterial or venous thrombosis;
2. To determine the dose of bivalirudin required to achieve adequate anticoagulation as measured by the activated clotting time (ACT) or activated partial thromboplastin time (aPTT) in Infants Under Six Months with arterial or venous thrombosis;
3. To determine the outcome of patients on bivalirudin with respect to thrombus resolution and bleeding complications compared to patients on unfractionated heparin (UH) or low molecular weight heparin (LMWH).

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal-guardian has provided written informed consent before initiation of any study related procedures.
* Objectively confirmed thrombotic event by either doppler ultrasound, echocardiogram, CT scan, MRI, MR angiogram, MR venogram, venogram or arteriogram.
* Age less than 6 months .
* Gestational age greater than 35 weeks
* Expected life expectancy at least 14 days.
* No contraindication to anticoagulation i.e. bleeding complications.

Exclusion Criteria:

* Active or recent (less than 7 days) bleeding.
* Known allergy to Angiomax or hirudin, or known sensitivity to any component of the product.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment.
* Refusal to undergo blood transfusion should it become necessary.
* Any other disease or condition, which, in the judgment of the Investigator would place a patient at undue risk by being enrolled in the trial.
* Baseline prolonged PT (>18 secs) or aPTT (>55 secs)
* Platelet count < 50,000 cells/mm3
* Birth Trauma
* Planned or indicated surgery within 30 days
* Major or minor bleeding event

Ages: 0 Years to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25
Dates: Start 2002-08; Study Completion 2004-12

PRIMARY OUTCOMES:
Observation of improvement for thrombosis or by clinical exam such as: Decrease in size of thrombus, restoration of flow through an occluded vessel, decrease in diameter of extremity or head.

SECONDARY OUTCOMES:
In addition, efficacy will also be judged by demonstrating a decrease in the molecular markers of thrombin generation.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Young, MD, Principal Investigator — Children's Hospital Orange County
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States